CLINICAL TRIAL: NCT05590260
Title: Prevention of Iron Deficiency Anemia Post-delivery (PRIORITY Trial): A Randomized Controlled Trial of the Global Network for Women's and Children's Health Research
Brief Title: Prevention of Iron Deficiency Anemia Post-delivery
Acronym: PRIORITY
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Thomas Jefferson University (Other); University of North Carolina, Chapel Hill (Other); Kinshasa School of Public Health (Other); University of Alabama at Birmingham (Other); University Teaching Hospital, Lusaka, Zambia (Other); University of Colorado, Denver (Other); Institute of Nutrition of Central America and Panama (Other); University of Virginia (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Columbia University (Other); Aga Khan University (Other); Boston University (Other); Lata Medical Research Foundation, Nagpur (Other); Indiana University (Other); Moi University (Other); RTI International (Other); Bill and Melinda Gates Foundation (Other); KLE University Jawaharlal Nehru Medical College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP PRIORITY
Record Dates: First submitted 2022-09-29; First posted 2022-10-21 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Postpartum Anemia
Keywords: Postpartum anemia; Anemia; Postpartum; IV Iron; Iron Tablets; Iron; Pregnancy; Maternal; Infant; Hemaglobin
MeSH Terms: conditions — Anemia | interventions — Iron

STUDY DESIGN:
Intervention Model Description: Study participation will be individually randomized and allocated 1:1 to one of two arms stratified by site. A computer algorithm generated by the data coordinating center (DCC) will create the random assignment to one of the treatment arms based on randomly permuted block design with randomly varied block sizes. Randomization will be stratified based on delivery mode (Cesarean section vs. vaginal birth) and site. The block sizes will be known only by the Data Coordinating Center's personnel.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IV iron arm (Experimental): Which will result in receipt of a single-dose IV iron infusion between 6 and 48 hours after delivery and prior to discharge from the facility; folate tablets per local guidelines.
  Interventions: Drug: IV iron infusion
- Oral iron comparator arm (Active Comparator): Oral iron tablets (containing 60 mg of elemental iron (± folate as per local guidelines)) to be taken at a treatment dose of twice daily for 6 weeks.
  Interventions: Drug: Oral iron tablets

INTERVENTIONS:
Drug: IV iron infusion — single-dose IV iron infusion
  Arms: IV iron arm
Drug: Oral iron tablets — 60 mg of elemental iron
  Arms: Oral iron comparator arm

SUMMARY:
PRIORITY is designed as a 2-arm, randomized-controlled trial focused on postpartum women. The trial will recruit women who are diagnosed with moderate anemia based on a blood sample taken 6-48 hours after childbirth. A total of 4,800 eligible women, or 600 women per research site, will be consented and enrolled in the trial. The study hypothesizes that at 6 weeks post-delivery, prevalence of the non-anemic state in women in that received a single-dose IV iron infusion between 6 and 48 hours after delivery and prior to discharge from the facility will be greater than that of women given a supply of oral iron tablets taken twice daily for 6 weeks.

DETAILED DESCRIPTION:
PRIORITY is a 2-arm, randomized-controlled trial (RCT) that will be implemented at 8 sites in 7 countries: Bangladesh, Democratic Republic of the Congo, Guatemala, India (Nagpur and Belagavi), Kenya, Pakistan, and Zambia. The research team for each site will enroll approximately 600 women who deliver at a hospital or other facility such as a health center with delivery services. Participants will be randomized to receive a single-dose IV iron infusion between 6 and 48 hours after delivery prior to discharge from the facility or oral iron tablets taken twice daily for 6 weeks. They will then be assessed by research staff at an appropriate health facility at 6 weeks and 6 months post-delivery by providing a maternal blood sample that will be analyzed to determine Hb concentration. At each study visit, trained staff will also measure serum ferritin, serum transferrin receptor, C-reactive protein (CRP) and alpha 1 acid glycoprotein (AGP). Additionally, in the African research sites, a rapid diagnostic test (RDT) for malaria will be administered upon admission to the birthing facility, and at 6 weeks and 6 months postpartum. The Edinburgh Postnatal Depression Scale (EPDS), The World Health Organization Quality-of-Life (QOL) scale, The Maternal Fatigue Severity Scale (FSS-5R), and The Mother-to-infant Bonding Scale (MIBS) will also be used at the 6 weeks and 6 months postpartum follow up appointments to collect data for secondary study aims.The study hypothesizes that at 6 weeks post-delivery, the prevalence of the non-anemic state in women in that received a single-dose IV iron infusion between 6 and 48 hours after delivery and prior to discharge from the facility will be greater than that of women given a supply of oral iron tablets taken twice daily for 6 weeks. Secondary study aims will look at the effects of postpartum depression on maternal quality of life, fatigue, and breastfeeding initiation and retention rates. Depression is also a risk factor for reducing infant-mother bonding.

The PRIORITY RCT will include an implementation research (IR) sub-study to complement the findings of the RCT trial and provide evidence about facilitators, barriers, and costs of implementation to inform global guidelines on the use of IV iron in postpartum women in Low-Middle Income Countries (LMIC). This Implementation Research (IR) sub-study will build upon the PRIORITY trial as well as other research projects to assess IV iron that are being conducted by the Jawaharlal Nehru Medical College research team in Belagavi, India, Thomas Jefferson University (TJU) and by the Aga Khan University team in Pakistan. The IR will utilize a mixed methods approach, employing both quantitative and qualitative data collection to better understand the potential barriers and facilitators to IV iron use in India and Pakistan. The implementation research will be harmonized with the timeline of the main PRIORITY trial, enabling the investigators to collect the IR data in parallel with the trial. The mixed methods IR study for the PRIORITY trial in India and Pakistan will be guided by the Consolidated Framework for Implementation Research (CFIR) and by Proctor's implementation outcomes framework. CFIR and Proctor's framework are complementary and provide a structure for guiding the types of questions and target groups for the implementation research data collection during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Established pregnancy >20 weeks gestation by LMP and/or clinical assessment and/ Or USG
* Age: 15 years (or lower limit age eligible*) to 49 years
* Confirmed moderate anemia (Hb 7.0 to 9.9 g/dL, 6-48 hour after delivery based on a venous blood sample on Hemocue®)
* Deliver in participating study hospital or health facility
* Able to provide informed consent
* Plans to remain in study area for duration of the study

Exclusion Criteria:

* IV Iron infusion received in past 3 weeks
* Contraindication to iron supplementation (some examples may include hemolytic anemia, allergy, severe infection)
* Blood transfusion already received or scheduled during the current hospital admission
* Known diagnosis of pre-existing depression or other psychiatric illness
* Stillbirth, major congenital anomaly, or neonatal loss prior to randomization
* Women testing positive and previously untreated for malaria
* Presenting with symptomatic anemia with dyspnea or fatigue and need for immediate correction
* Women with known hemoglobinopathy (sickle cell disease or thalassemia)
* Presence of severe allergic conditions such as severe asthma or known drug allergies
* Women presenting with any illness/condition requiring immediate medical care per physician's assessment

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4800 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of women with non-anemic hemaglobin levels (Hb >11 g/dL) | 6 weeks post-delivery
  Hemoglobin measure

SECONDARY OUTCOMES:
Number of maternal deaths | From delivery to 6 months post-delivery
  Maternal death from any cause
Number of women who receive a blood transfusion post-discharge | through 6 months post-delivery
  Blood transfusion given to mother enrolled in study after randomization
Number of women who experience a postpartum hemorrhage requiring transfusion or major surgery | from intervention through 6 weeks post-delivery
  Postpartum hemorrhaging defined as those requiring transfusion of surgery
Number of women with hospitalization | through 6 months post-delivery
  Hospital admission for any reason after randomization until 6 months postpartum
Number of women with documentation of postpartum complications | Randomization through 6 weeks post delivery
  Maternal postpartum clinical complications
Number of women screening positive for postpartum depression | 6 weeks and 6 months
  Edinburgh Postnatal Depression Scale (EPDS) will be used as post-partum depression screening tool
Number of women with severe fatigue | 6 weeks and 6 months
  Fatigue severity score (utilizing 9 question survey with a scale from 1-7 for each item; the lower the total score is the better the outcome)
Differences between treatment groups in infant-mother bonding scale scores | 6 weeks
  Will utilize mother-infant (MIBS) tool
Differences in quality of life assessment scores | 6 weeks and 6 months
  Will utilize WHO Quality of Life (QOL) - BREF tool. The minimum is 0 (bad QOL) and maximum is 100 (good QOL).
Prevalence of severe/moderate/mild anemia among women | 6 weeks and 6 months
  Use Hemocue hemoglobin measure to categorize anemia
Maternal - Change resulting in severe/moderate/mild anemia by treatment arm | 6 months
  Evaluate individual changes in maternal anemia levels from randomization to 6 months
Maternal - Hemoglobin concentration by mode of delivery | 6 months
  Evaluate hemoglobin stratified by Cesarean delivery vs. Vaginal delivery
Maternal - Differences in ferritin and inflammatory markers by treatment group | 6 weeks, 6 months
  Using centralized testing, evaluate differences by treatment group
Number of neonatal infant deaths | birth to 6 months
  Neonatal or infant death from any cause post-randomization
Number of infants with hospitalization | birth to 6 months
  Neonatal or infant hospitalization for any reason
Number of women exclusive breastfeeding rate and intend to continue breastfeeding through 12 months post-delivery | 6 weeks and 6 months
  Self report of breastfeeding

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Derman, MD, MPH, Principal Investigator — Thomas Jefferson University, Philadelphia, PA
Locations (8):
- ICDDRB, Dhaka, Bangladesh
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo
- INCAP, Guatemala City, Guatemala
- India (2):
  - KLE Society's Jawaharlal Nehru Medical College, Belagavi, Karnataka
  - Lata Medical Research Foundation, Nagpur
- Moi University School of Medicine, Eldoret, Kenya
- The Aga Khan University, Karachi, Pakistan
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sultan P, Bampoe S, Shah R, Guo N, Estes J, Stave C, Goodnough LT, Halpern S, Butwick AJ. Oral vs intravenous iron therapy for postpartum anemia: a systematic review and meta-analysis. Am J Obstet Gynecol. 2019 Jul;221(1):19-29.e3. doi: 10.1016/j.ajog.2018.12.016. Epub 2018 Dec 19. PMID 30578747
- [Background] Matsunaga A, Ohashi Y, Sakanashi K, Kitamura T. Factor structure of the Postpartum Bonding Questionnaire: Configural invariance and measurement invariance across postpartum time periods. J Psychiatr Res. 2021 Mar;135:1-7. doi: 10.1016/j.jpsychires.2020.11.017. Epub 2020 Nov 9. PMID 33388520
- [Background] Taylor A, Atkins R, Kumar R, Adams D, Glover V. A new Mother-to-Infant Bonding Scale: links with early maternal mood. Arch Womens Ment Health. 2005 May;8(1):45-51. doi: 10.1007/s00737-005-0074-z. Epub 2005 May 4. PMID 15868385
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Fellmeth G, Harrison S, Opondo C, Nair M, Kurinczuk JJ, Alderdice F. Validated screening tools to identify common mental disorders in perinatal and postpartum women in India: a systematic review and meta-analysis. BMC Psychiatry. 2021 Apr 20;21(1):200. doi: 10.1186/s12888-021-03190-6. PMID 33879130
- [Background] Shrestha SD, Pradhan R, Tran TD, Gualano RC, Fisher JR. Reliability and validity of the Edinburgh Postnatal Depression Scale (EPDS) for detecting perinatal common mental disorders (PCMDs) among women in low-and lower-middle-income countries: a systematic review. BMC Pregnancy Childbirth. 2016 Apr 4;16:72. doi: 10.1186/s12884-016-0859-2. PMID 27044437
- [Background] Ali SA, Tikmani SS, Saleem S, Patel AB, Hibberd PL, Goudar SS, Dhaded S, Derman RJ, Moore JL, McClure EM, Goldenberg RL. Hemoglobin concentrations and adverse birth outcomes in South Asian pregnant women: findings from a prospective Maternal and Neonatal Health Registry. Reprod Health. 2020 Nov 30;17(Suppl 2):154. doi: 10.1186/s12978-020-01006-6. PMID 33256770
- [Background] Jessani S, Saleem S, Hoffman MK, Goudar SS, Derman RJ, Moore JL, Garces A, Figueroa L, Krebs NF, Okitawutshu J, Tshefu A, Bose CL, Mwenechanya M, Chomba E, Carlo WA, Das PK, Patel A, Hibberd PL, Esamai F, Liechty EA, Bucher S, Nolen TL, Koso-Thomas M, Miodovnik M, McClure EM, Goldenberg RL. Association of haemoglobin levels in the first trimester and at 26-30 weeks with fetal and neonatal outcomes: a secondary analysis of the Global Network for Women's and Children's Health's ASPIRIN Trial. BJOG. 2021 Aug;128(9):1487-1496. doi: 10.1111/1471-0528.16676. Epub 2021 Apr 12. PMID 33629490
- [Background] Parks S, Hoffman MK, Goudar SS, Patel A, Saleem S, Ali SA, Goldenberg RL, Hibberd PL, Moore J, Wallace D, McClure EM, Derman RJ. Maternal anaemia and maternal, fetal, and neonatal outcomes in a prospective cohort study in India and Pakistan. BJOG. 2019 May;126(6):737-743. doi: 10.1111/1471-0528.15585. Epub 2019 Jan 24. PMID 30554474
- [Background] Patel A, Prakash AA, Das PK, Gupta S, Pusdekar YV, Hibberd PL. Maternal anemia and underweight as determinants of pregnancy outcomes: cohort study in eastern rural Maharashtra, India. BMJ Open. 2018 Aug 8;8(8):e021623. doi: 10.1136/bmjopen-2018-021623. PMID 30093518
- [Background] Rioux FM, Savoie N, Allard J. Is there a link between postpartum anemia and discontinuation of breastfeeding? Can J Diet Pract Res. 2006 Summer;67(2):72-6. doi: 10.3148/67.2.2006.72. PMID 16759433
- [Background] Babu GR, Murthy GVS, Singh N, Nath A, Rathnaiah M, Saldanha N, Deepa R, Kinra S. Sociodemographic and Medical Risk Factors Associated With Antepartum Depression. Front Public Health. 2018 May 2;6:127. doi: 10.3389/fpubh.2018.00127. eCollection 2018. PMID 29770322
- [Background] Tsai AC, Scott JA, Hung KJ, Zhu JQ, Matthews LT, Psaros C, Tomlinson M. Reliability and validity of instruments for assessing perinatal depression in African settings: systematic review and meta-analysis. PLoS One. 2013 Dec 10;8(12):e82521. doi: 10.1371/journal.pone.0082521. eCollection 2013. PMID 24340036
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Khaskheli MN, Baloch S, Sheeba A, Baloch S, Khaskheli FK. Iron deficiency anaemia is still a major killer of pregnant women. Pak J Med Sci. 2016 May-Jun;32(3):630-4. doi: 10.12669/pjms.323.9557. PMID 27375704
- [Background] Kramer MS, Dahhou M, Vallerand D, Liston R, Joseph KS. Risk factors for postpartum hemorrhage: can we explain the recent temporal increase? J Obstet Gynaecol Can. 2011 Aug;33(8):810-819. doi: 10.1016/S1701-2163(16)34984-2. PMID 21846436
- [Background] Markova V, Norgaard A, Jorgensen KJ, Langhoff-Roos J. Treatment for women with postpartum iron deficiency anaemia. Cochrane Database Syst Rev. 2015 Aug 13;2015(8):CD010861. doi: 10.1002/14651858.CD010861.pub2. PMID 26270434
- [Background] Vanobberghen F, Lweno O, Kuemmerle A, Mwebi KD, Asilia P, Issa A, Simon B, Mswata S, Schmidlin S, Glass TR, Abdulla S, Daubenberger C, Tanner M, Meyer-Monard S. Efficacy and safety of intravenous ferric carboxymaltose compared with oral iron for the treatment of iron deficiency anaemia in women after childbirth in Tanzania: a parallel-group, open-label, randomised controlled phase 3 trial. Lancet Glob Health. 2021 Feb;9(2):e189-e198. doi: 10.1016/S2214-109X(20)30448-4. Epub 2020 Nov 24. PMID 33245866
- [Background] Skevington SM. Measuring quality of life in Britain: introducing the WHOQOL-100. J Psychosom Res. 1999 Nov;47(5):449-59. doi: 10.1016/s0022-3999(99)00051-3. PMID 10624843
- [Background] Young CA, Mills R, Al-Chalabi A, Burke G, Chandran S, Dick DJ, Ealing J, Hanemann CO, Harrower T, Mcdermott CJ, Majeed T, Pinto A, Talbot K, Walsh J, Williams TL, Tennant A; TONiC study group. Measuring quality of life in ALS/MND: validation of the WHOQOL-BREF. Amyotroph Lateral Scler Frontotemporal Degener. 2020 Jun 27;21(5-6):364-372. doi: 10.1080/21678421.2020.1752244. PMID 32597226
- [Background] Auerbach M, Macdougall I. The available intravenous iron formulations: History, efficacy, and toxicology. Hemodial Int. 2017 Jun;21 Suppl 1:S83-S92. doi: 10.1111/hdi.12560. Epub 2017 Mar 29. PMID 28371203
- [Background] Chertow GM, Mason PD, Vaage-Nilsen O, Ahlmen J. Update on adverse drug events associated with parenteral iron. Nephrol Dial Transplant. 2006 Feb;21(2):378-82. doi: 10.1093/ndt/gfi253. Epub 2005 Nov 11. PMID 16286429
- [Background] Gomez-Ramirez S, Shander A, Spahn DR, Auerbach M, Liumbruno GM, Vaglio S, Munoz M. Prevention and management of acute reactions to intravenous iron in surgical patients. Blood Transfus. 2019 Mar;17(2):137-145. doi: 10.2450/2018.0156-18. Epub 2018 Oct 16. PMID 30418128
- [Background] Rampton D, Folkersen J, Fishbane S, Hedenus M, Howaldt S, Locatelli F, Patni S, Szebeni J, Weiss G. Hypersensitivity reactions to intravenous iron: guidance for risk minimization and management. Haematologica. 2014 Nov;99(11):1671-6. doi: 10.3324/haematol.2014.111492. PMID 25420283
- [Background] Tolkien Z, Stecher L, Mander AP, Pereira DI, Powell JJ. Ferrous sulfate supplementation causes significant gastrointestinal side-effects in adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 20;10(2):e0117383. doi: 10.1371/journal.pone.0117383. eCollection 2015. PMID 25700159
- [Background] Auerbach M, Macdougall IC. Safety of intravenous iron formulations: facts and folklore. Blood Transfus. 2014 Jul;12(3):296-300. doi: 10.2450/2014.0094-14. No abstract available. PMID 25074787
- [Background] Rebecca Giallo, Catherine Wade & Mandy Kienhuis (2014) Fatigue in mothers of infants and young children: factor structure of the fatigue assessment scale, Fatigue: Biomedicine, Health & Behavior, 2:3, 119-131, DOI: 10.1080/21641846.2014.925326
- See also: Auerbach M. Treatment of iron deficiency anemia in adults. 2020 — http://www.uptodate.com/contents/treatment-of-iron-deficiency-anemia-in-adults
- See also: Electronic Medicines Compendium (eMC). Monofer 100mg/ml solution for injection/infusion. — http://www.medicines.org.uk/emc/product/5676/smpc
- See also: Electronic Medicines Compendium (eMC). Ferinject (ferric carboxymaltose). — http://www.medicines.org.uk/emc/product/5910/smpc
- See also: World Health Organization. Anemia — http://www.who.int/health-topics/anaemia
- See also: World Health Organization. Maternal health — http://www.who.int/health-topics/maternal-health
- See also: World Health Organization. Prevalence of anaemia in women of reproductive age (aged 15-49) (%) — http://www.who.int/data/gho/data/indicators/indicator-details/GHO/prevalence-of-anaemia-in-women-of-reproductive-age-(-)
- See also: World Health Organization. The World Health Organization Quality of Life (WHOQOL). 2012. — http://www.who.int/publications/i/item/WHO-HIS-HSI-Rev.2012.03
- See also: World Health Organization. WHA65.6. Comprehensive implementation plan on maternal, infant and young child nutrition as passed by the World Health Assembly at the Sixty-fifth World Health Assembly meeting.2012. — http://apps.who.int/iris/bitstream/handle/10665/113048/WHO_NMH_NHD_14.1_eng.pdf;jsessionid=639F57F1C9B591D01291EECF0D9E632A?sequence=1